CLINICAL TRIAL: NCT02301923
Title: Predictive Factors Determining Continuous Positive Airway Pressure (CPAP) Compliance in Obstructive Sleep Apnea
Brief Title: Continuous Positive Airway Pressure (CPAP) Compliance in Obstructive Sleep Apnea
Acronym: CPAPcompl
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Saint-Joseph University (Other)
Responsible Party: Principal Investigator, May Samaha, Moussa Riachy MD FCCP, Saint-Joseph University
Other Study IDs: HDF575
Record Dates: First submitted 2014-11-02; First posted 2014-11-26 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Sleep Apnea, Obstructive; Patient Compliance
Keywords: Continuous Positive Airway Pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- CPAP compliant (C): Patients confirmed with obstructive sleep apnea and succeeded to pursue treatment with CPAP
- CPAP noncompliant (NC): Patients confirmed with obstructive sleep apnea but did not succeed to pursue treatment with CPAP

SUMMARY:
This study aims to determine the average compliance of a patient under CPAP therapy for obstructive sleep apnea as well as the various factors that influence it.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea (OSA) is a frequent disease that affects 4% of the male population and 2% of the female population, with well known repercussions on the quality of life (daytime drowsiness, concentration issues, increased motor vehicle accidents, etc) and cardiovascular risk (increased risk of strokes, hypertension, diabetes, CAD, etc.). It is caused by an intermittent relaxation of the throat muscles during sleep, thus blocking the airways and leading to snoring and apnea.

Treatment can involve diets and sports, sleep hygiene techniques, mandibular advancement devices. But the CPAP (continuous positive airway pressure) device remains the first line therapy for OSA. It is very effective at reducing apnea-hypopnea (AHI) and oxygen desaturation indexes (ODI), but poor compliance is often noticed, with only 46% of patients still using the device at 6 months.

Despite numerous studies on the subject, very few have included a large number of patients(>150) or long follow up time (>1 year), or reached conclusive evidence concerning the factors that influence CPAP compliance.

In order to determine these factors, the investigators have taken into account approximately 450 patients over a timeframe of 5 years who have used a CPAP device during the course of their disorder, and established a Kaplan-Meyer estimation of their survival function. The investigators have then used anthropometry (BMI, neck circumference, sex, age, etc.), polysomnography (Epworth score, AHI, ODI, sleep efficiency, etc.) and CPAP (pressures, leaks, etc.) data with a Cox regression in order to determine the factors that influence the compliance of a patient.

The results will allow us to establish the average compliance of a patient under CPAP therapy, as well as the reasons leading to its termination, the factors predicting a decreased compliance and the consequences of stopping the treatment. This will allow us to set up multiple methods of improved follow-up in patients that are predicted recalcitrant to CPAP therapy.

ELIGIBILITY:
Inclusion Criteria:

* All HDF patients with OSA, treated for at least one day by CPAP, from the period of June 2008 to June 2013.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with OSA in the sleep center of Hotel Dieu de France (HDF) hospital, treated for at least one day by CPAP, from the period of June 2008 to June 2013.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2014-11; Primary Completion 2014-11 (Actual); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Compliance time to CPAP | 6 years
  Survival study taking the noncompliance to CPAP treatment as an event

SECONDARY OUTCOMES:
Predictive factors related to the patient for compliance to CPAP (Sociologic and economic status, medical co morbidities, Anthropometric characteristics) | 6 years
  Factors related to the patient: Sociologic and economic status, medical co morbidities, Anthropometric characteristics.
Predictive factors related to the provider for compliance to CPAP (Attitude of the provider (active, passive), consistency/quality of the follow up) | 6 years
  Factors related to the provider: Attitude of the provider (active, passive), consistency/quality of the follow up.
Predictive factors related to the device for compliance to CPAP (Mask type, use of a humidification, Device type/mode, Pressure set, Cost, Side effects) | 6 years
  Factors related to the device: Mask type, use of a humidification, Device type/mode, Pressure set, Cost, Side effects.
Predictive factors related to OSA for compliance to CPAP (Severity score, fatigue and Epworth score, Polysomnography profile (AHI, ODI, Arousal index…), use of alternative treatments) | 6 years
  Factors related to OSA: Severity score, fatigue and Epworth score, Polysomnography profile (AHI, ODI, Arousal index…), use of alternative treatments.
Cardiovascular outcome/benefits (cardiovascular events; defined by hypertension, coronary event, stroke, diabetes, cardiac insufficiency, arrhythmias) | 6 years
  cardiovascular events; defined by hypertension, coronary event, stroke, diabetes, cardiac insufficiency, arrhythmias; timeframe: after CPAP cessation

CONTACTS AND LOCATIONS:
Overall Officials: Moussa Riachy, Ass Prof, Principal Investigator — Saint Joseph Univ
Locations (1):
- Hotel Dieu de France Hospital, Beirut, Lebanon

REFERENCES:
- See also: Bibliography — https://drive.google.com/drive/#folders/0B4QQ7AWZ3tQ2a2tnZlp4MGpoLU0/0B7PwtSh2G1XgTWJmRFowQlA0YWM